CLINICAL TRIAL: NCT04091737
Title: A Phase 1 Pilot Study to Evaluate the Safety and Feasibility of Gene Therapy With CSL200 (Autologous Enriched CD34+ Cell Fraction That Contains CD34+ Cells Transduced With Lentiviral Vector Encoding Human γ-GlobinG16D and Short-Hairpin RNA734) in Adult Subjects With Severe Sickle Cell Disease
Brief Title: CSL200 Gene Therapy in Adults With Severe Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unanticipated delays, not for safety reasons
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL200_1001
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CSL200 (Experimental): Autologous enriched CD34+ cell fraction that contains CD34+ cells transduced with lentiviral vector encoding human γ-globinG16D and short-hairpin RNA734
  Interventions: Biological: Autologous enriched CD34+ cell fraction that contains CD34+ cells transduced with lentiviral vector encoding human γ-globinG16D and short-hairpin RNA734

INTERVENTIONS:
Biological: Autologous enriched CD34+ cell fraction that contains CD34+ cells transduced with lentiviral vector encoding human γ-globinG16D and short-hairpin RNA734 — * Cryopreserved formulated autologous enriched CD34+ cell fraction that contains CD34+ cells transduced with lentiviral vector encoding human γ-globinG16D and short-hairpin RNA734 in a bag for infusion
  * Plerixafor to mobilize hematopoietic stem cells prior to each apheresis
  * Single dose melphalan before administration of CSL200
  Other Names: CSL200

SUMMARY:
This is a phase 1 pilot study of CSL200 in adult subjects with severe sickle cell disease. The primary objectives of this study are to evaluate the safety of the following: collection of CD34+ hematopoietic stem / progenitor cells by apheresis after mobilization with plerixafor, reduced intensity conditioning with melphalan, and administration of CSL200.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease with the homozygous HbS homozygous genotype (HbSS) or an HbSβ thalassemia variant (ie, HbSβ0 thalassemia or HbSβ+ thalassemia) genotype, confirmed by hemoglobin studies.
* Fetal hemoglobin (HbF) ≤ 15%.
* Severe sickle cell disease symptomatology, defined as any one or more of the following:

  1. ≥ 2 episodes of acute chest syndrome in the last 2 years.
  2. ≥ 3 episodes of severe pain events requiring a visit to a medical facility and treatment with opioids in the last 2 years.
  3. > 2 episodes of recurrent priapism in the last 2 years.
  4. Red-cell alloimmunization (> 2 antibodies) during long-term transfusion therapy (lifetime history).
  5. Chronic transfusions for primary or secondary prophylaxis (lifetime history).
  6. Trans-thoracic echocardiograph evidence of tricuspid valve regurgitant jet velocity ≥ 2.7 m/sec (lifetime history).
  7. Clinically significant neurologic event (eg, ischemic stroke) or any neurological deficit lasting > 24 hours.
* Not eligible for human leukocyte antigen (HLA)-matched hematopoietic stem cell transplantation, defined as follows: no medically eligible, available, and willing 10/10 matched HLA-identical sibling donor, unless subject has declined this treatment option (as documented in the informed consent form).
* Not eligible for, declined, or, as judged by the investigator, failed therapy with hydroxyurea and if still on hydroxyurea is able to interrupt hydroxyurea starting at the beginning of the transfusions, before mobilization and apheresis.

Exclusion Criteria:

* Hypoxanthine-guanine phosphoribosyl transferase (HPRT) deficiency.
* Thiopurine S-methyltransferase (TPMT) deficiency.
* Alpha thalassemia.
* Inadequate bone marrow function, defined as at least 1 of the following:

  1. Absolute neutrophil count < 1000/µL.
  2. Platelet count < 120,000/µL.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) associated with the administration of CSL200 | Up to 48 weeks
  Adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
  Serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is medically significant.
  Adverse event of special interest (AESI) is defined in this study as any of the following: acute immune reactions, autoimmunity to CSL200; malignancy; predominant integration site in presence of malignancy or other abnormality.
Number of subjects experiencing AEs, SAEs, and AESIs associated with the administration of CSL200 | Up to 48 weeks
Number of AEs, SAEs, and AESIs associated with the collection of CD34+ HSPCs by apheresis after mobilization with plerixafor | Up to 6 weeks
Number of subjects experiencing AEs, SAEs, and AESIs associated with the collection of CD34+ HSPCs by apheresis after mobilization with plerixafor | Up to 6 weeks
Number of AEs, SAEs, and AESIs associated with reduced intensity conditioning with melphalan | Up to 3 weeks
Number of subjects experiencing AEs, SAEs, and AESIs associated with reduced intensity conditioning with melphalan | Up to 3 weeks

SECONDARY OUTCOMES:
Total by-subject number of CD34+ HSPCs collected in total and in each apheresis session | Up to 2 days
  Collection of CD34+ HSPCs by apheresis after mobilization with plerixafor assessed by CD34+ HSPCs collected
Number of subjects receiving plerixafor and number of plerixafor doses administered by subject | Up to 2 days
  Collection of CD34+ HSPCs by apheresis after mobilization with plerixafor assessed by plerixafor administrations
Number of subjects undergoing apheresis and number of apheresis sessions by subject | Up to 2 days
  Collection of CD34+ HSPCs by apheresis after mobilization with plerixafor assessed by apheresis sessions
The number of subjects undergoing reduced intensity conditioning with melphalan and able to receive CSL200 | 2 days
  Reduced intensity conditioning assessed by subjects receiving melphalan
Number of subjects receiving CSL200 | 1 day
By-subject number of separate CSL200 drug products administered | 1 day
Number of CSL200 CD34+ HSPCs/kg administered by subject and by CSL200 drug product | 1 day
By-subject total number and percentage of CD34+ HSPCs transduced with CAL-H | Up to 48 weeks
Vector copy number (VCN) | Up to 48 weeks
  VCN will be determined by using the average number of CAL-H vector genomes per cell

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.